CLINICAL TRIAL: NCT00912418
Title: Pilot Study for the Evaluation of the Efficacy of Vaccination With Autologous Tumor Cells Plus GM-CSF-in-adjuvant, Followed by Systemic Low-dose-IL-2 Administration, in Patients With High Risk Melanoma.
Brief Title: Pilot Study for the Evaluation of the Efficacy of Vaccination With Autologous Tumor Cells Plus Granulocyte-macrophage Colony-stimulating Factor (GM-CSF) - in - Adjuvant, Followed by Systemic Low-dose-interleukin-2 (IL-2) Administration, in Patients With High Risk Melanoma
Acronym: MEL37
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Craig L Slingluff, Jr (Other)
Responsible Party: Sponsor-Investigator, Craig L Slingluff, Jr, Director, Human Immune Therapy Center, University of Virginia
Organization: University of Virginia (Other)
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8577
Record Dates: First submitted 2009-06-01; First posted 2009-06-03 (Estimated); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Melanoma
Keywords: melanoma; vaccine; IL2 low dose
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: autologous tumor cells plus GM-CSF-in Adjuvant — Autologous tumor cells plus 225 ug GM-CSF in-adjuvant: The autologous tumor cells will be administered intradermally. Subjects will be vaccinated over at least a 6 week period (at weeks 0, 1, 2, 4, 5, 6), with responders vaccinated every 4 weeks thereafter for a maximum of 9 vaccinations (up to week 18). Systemic low-dose interleukin-2 will also be administered daily for 6 weeks following the second vaccination at week 1.
  Concurrent with the first three of these vaccinations, each patient will also receive an additional set of 3 vaccinations in a different site, the response to which will be evaluated at the draining lymph node. This node will be harvested using lymphatic mapping and sentinel node biopsy methods.

SUMMARY:
This study is an open-label, pilot study of an autologous tumor cell vaccine.

DETAILED DESCRIPTION:
Regimen: A vaccine comprising autologous melanoma cells plus GM-CSF in-adjuvant will be administered intradermally at a single dose. Subjects will be vaccinated over at least a 6 week period (at weeks 0, 1, 2, 4, 5, 6), with responders vaccinated every 4 weeks thereafter for a maximum of 9 vaccinations (up to week 18). Systemic low-dose interleukin-2 will also be administered daily for 6 weeks following the second vaccination at week 1.

Concurrent with the first three of these vaccinations, each patient will also receive an additional set of 3 vaccinations in a different site, the response to which will be evaluated at the draining lymph node. This node will be harvested using lymphatic mapping and sentinel node biopsy methods.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been diagnosed, by cytologic or histologic examination, with stage III or stage IV melanoma, where sufficient resected tumor is available for vaccine preparation (approximately 3 g tumor).
* Measurable tumor after resection is not required.
* Patients with up to 3 brain metastases may be included if the metastases are all < 2 cm in diameter, are asymptomatic, and there is no mass effect or they have been treated successfully by surgical excision or by gamma knife radiation therapy.
* Patients who have had a larger number of brain metastases resected or treated and resolved after gamma knife radiation therapy may be included if their status at the time of study initiation meets these criteria.
* For those patients with resected melanoma, surgical resections must have been performed within 6 months prior to entry. All patients must have:

  * ECOG performance status 0-1, and, ability and willingness to give informed consent.
  * Laboratory parameters as follows: ANC > 1000/mm3, and Platelets > 100,000 and Hgb > 10.
  * Hepatic: AST and ALT up to 1.5 x upper limits of normal (ULN), Bilirubin within ULN, Alkaline phosphatase up to 1.5 x ULN
  * Renal: Creatinine within ULN
  * Serology: HIV negative, Hepatitis C virus-negative.
* Patients who are not candidates for interferon, for people who decide not to take interferon, or for people who have failed interferon therapy (those patients who have progressed while on interferon therapy or who experienced a major toxicity while receiving treatment).

Exclusion Criteria:

* Patients who are currently receiving cytotoxic chemotherapy or radiation therapy, or who have received that therapy within the preceding 4 weeks.
* Patients who are currently receiving investigational agents, or who have received investigational agents within the preceding 30 days.
* Patients with known or suspected allergies to any component of the vaccine.
* Patients receiving the following medications at study entry or within 30 days are excluded:

  * Allergy desensitization injections
  * Corticosteroids, administered parenterally or orally.
* Topical corticosteroids are acceptable, Any growth factors, Interferons, Interleukin 2 (IL-2).
* Prior melanoma vaccinations will not be an exclusion criteria if given more than 8 weeks previously, but will be recorded, and data analysis will take this into account.
* Other investigational drugs or investigational therapy also will not necessarily be an exclusion criteria, but will similarly be recorded and taken into account during data analysis.
* Pregnancy or the possibility of becoming pregnant during vaccine administration.
* Female patients of child-bearing potential must have a negative pregnancy test (urinary or serum beta-HCG) prior to administration of the first vaccine dose.
* Males and females must agree, in the consent form, to use effective birth control methods during the course of vaccination. This is consistent with existing standards of practice for vaccine and chemotherapy protocols.
* Patients in whom there is a medical contraindication or other potential medical problem in complying with the requirements of the protocol, in the opinion of the investigator.
* Patients classified according to the New York Heart Association classification system as having Class II, III or IV heart disease.
* Patients with active connective tissue disease requiring medications, or other severe autoimmune disease.
* Patients who are actively hyperthyroid.
* Patients with uncontrolled diabetes.
* Patients with known allergies to penicillin, streptomycin, and amphotericin B.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2000-05-01 (Actual); Primary Completion 2002-09-17 (Actual); Study Completion 2002-10-09 (Actual)

PRIMARY OUTCOMES:
Cytotoxic T-cell response to autologous tumor (as measured by staining assay)

SECONDARY OUTCOMES:
Cytotoxic T-cell response to defined melanoma antigens. 1: Activation antigen expression by lymph node T-cells 2: Delayed-type hypersensitivity response to autologous tumor cells. 3: Antibody response to autologous tumor cells.

CONTACTS AND LOCATIONS:
Overall Officials: Craig L Slingluff, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States